CLINICAL TRIAL: NCT04442854
Title: A Randomized Controlled Trial of Cognitive Behavioral Group Prevention Program for Mainland Chinese University Students in Hong Kong
Brief Title: Cognitive Behavioral Group Therapy for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Jiayan Pan, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12607815
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Cognitive Behavior Group Therapy
Keywords: Chinese university student; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive behavioral group therapy (Experimental): A cognitive behavioral group prevention program An 8-session, cognitive behavioral group prevention program, featuring cultural appropriateness. One session per week, 3 hours for each session. The program contents include psychoeducation, cognitive skills training to identify and challenge maladaptive cognitions, and behavioral skills training. Each session contains mood check and homework. Participants' own examples are used in the group to demonstrate the CBT skills.
  Interventions: Other: cognitive behavioral group therapy
- Wait-list control group (No Intervention): No immediate intervention No intervention was provided when the experimental group was receiving services, but the same cognitive behavioral group prevention program was delivered to the wait-list control group after that.

INTERVENTIONS:
Other: cognitive behavioral group therapy — A 8-session cognitive behavior group intervention tailor-made for Mainland Chinese university students in Hong Kong
  Arms: cognitive behavioral group therapy

SUMMARY:
This study developed a culturally appropriate cognitive behavioral group prevention program for Mainland Chinese university students in Hong Kong. The effects of the group prevention program on psychological distress, acculturative stress, cognitions, emotions, and post-migration growth were examined.

DETAILED DESCRIPTION:
Detailed description:

Previous research has found the effectiveness of group cognitive behavioral therapy in improving international students' mental health and facilitating their psychological adaptation. However, this kind of research in Chinese societies is scant and previous studies lack control group in study design. This study developed an 8-session culturally appropriate cognitive behavioral group prevention program for Mainland Chinese university students in Hong Kong. Research design of randomized controlled trial was adopted. Program effectiveness was evaluated at both cognitive and emotional levels, including psychological distress, acculturative stress, emotions, automatic thoughts, sense-making coping, core belief re-examination and post-migration growth.

ELIGIBILITY:
Inclusion Criteria:

* Chinese students from Mainland China who were studying at local universities in Hong Kong
* GHQ-12 score of 2 or above (0-0-1-1)
* Willingness to participate in the study

Exclusion Criteria:

* GHQ-12 score of 11 or above (0-0-1-1)
* One or more psychotic disorders
* Severe depression diagnosed by professionals with suicidal attempts/ideation in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire-12 (GHQ-12) | pre-test at intake interview
  12 item rating scale measuring psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 (GHQ-12) | post-test at the end of the last session of the CBT group (for the experimental group), and when the experimental group finished the intervention (for the waitlist control group), respectively.
  12 item rating scale measuring psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 (GHQ-12) | 3-month follow-up test three months after completing the intervention
  12 item rating scale measuring psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
Acculturative Stress Scale for Chinese Students (ASSCS) | pre-test at intake interview
  35-item rating scale measuring acculturative stress, scale score ranges from 0-3, with a higher score indicating a higher level of acculturative stress
Acculturative Stress Scale for Chinese Students (ASSCS) | post-test at the end of the last session of the CBT group (for the experimental group), and when the experimental group finished the intervention (for the waitlist control group), respectively.
  35-item rating scale measuring acculturative stress, scale score ranges from 0-3, with a higher score indicating a higher level of acculturative stress
Acculturative Stress Scale for Chinese Students (ASSCS) | 3-month follow-up test three months after completing the intervention
  35-item rating scale measuring acculturative stress, scale score ranges from 0-3, with a higher score indicating a higher level of acculturative stress

SECONDARY OUTCOMES:
Chinese Automatic Thoughts Questionnaire (CATQ) | pre-test at intake interview
  14-item rating scale measuring automatic thoughts, subscale score ranges from 1-5 for the positive thought subscale and negative thought subscale
Chinese Automatic Thoughts Questionnaire (CATQ) | post-test at the end of the last session of the CBT group (for the experimental group), and when the experimental group finished the intervention (for the waitlist control group), respectively.
  14-item rating scale measuring automatic thoughts, subscale score ranges from 1-5 for the positive thought subscale and negative thought subscale
Chinese Automatic Thoughts Questionnaire (CATQ) | 3-month follow-up test three months after completing the intervention
  14-item rating scale measuring automatic thoughts, subscale score ranges from 1-5 for the positive thought subscale and negative thought subscale
Post-migration Growth Scale (PMGS) | pre-test at intake interview
  14-item rating scale measuring personal growth after migration, scale score ranges from 1-6, with a higher score indicating a higher level of post-migration growth
Post-migration Growth Scale (PMGS) | post-test at the end of the last session of the CBT group (for the experimental group), and when the experimental group finished the intervention (for the waitlist control group), respectively.
  14-item rating scale measuring personal growth after migration, scale score ranges from 1-6, with a higher score indicating a higher level of post-migration growth
Post-migration Growth Scale (PMGS) | 3-month follow-up test three months after completing the intervention
  14-item rating scale measuring personal growth after migration, scale score ranges from 1-6, with a higher score indicating a higher level of post-migration growth
Chinese Making Sense of Adversity Scale (CMSAS) | pre-test at intake interview
  12-item rating scale measuring sense-making coping strategies of Chinese people, scale score ranges from 1-6, with higher scores indicating a greater tendency to use the sense-making coping
Chinese Making Sense of Adversity Scale (CMSAS) | post-test at the end of the last session of the CBT group (for the experimental group), and when the experimental group finished the intervention (for the waitlist control group), respectively.
  12-item rating scale measuring sense-making coping strategies of Chinese people, scale score ranges from 1-6, with higher scores indicating a greater tendency to use the sense-making coping
Chinese Making Sense of Adversity Scale (CMSAS) | 3-month follow-up test three months after completing the intervention
  12-item rating scale measuring sense-making coping strategies of Chinese people, scale score ranges from 1-6, with higher scores indicating a greater tendency to use the sense-making coping
Core Belief Inventory (CBI) | pre-test at intake interview
  9-item rating scale measuring core belief re-examination, scale score ranges from 0-5, with a higher score indicating a higher level of core belief re-examination
Core Belief Inventory (CBI) | post-test at the end of the last session of the CBT group (for the experimental group), and when the experimental group finished the intervention (for the waitlist control group), respectively.
  9-item rating scale measuring core belief re-examination, scale score ranges from 0-5, with a higher score indicating a higher level of core belief re-examination
Core Belief Inventory (CBI) | 3-month follow-up test three months after completing the intervention
  9-item rating scale measuring core belief re-examination, scale score ranges from 0-5, with a higher score indicating a higher level of core belief re-examination
Chinese Affect Scale (CAS) | pre-test at intake interview
  20-item rating scale measuring trait and state affect of Chinese-speaking people, subscale scores range from 1-6, with a higher score indicating a higher level of positive/negative emotion
Chinese Affect Scale (CAS) | post-test at the end of the last session of the CBT group (for the experimental group), and when the experimental group finished the intervention (for the waitlist control group), respectively.
  20-item rating scale measuring trait and state affect of Chinese-speaking people, subscale scores range from 1-6, with a higher score indicating a higher level of positive/negative emotion
Chinese Affect Scale (CAS) | 3-month follow-up test three months after completing the intervention
  20-item rating scale measuring trait and state affect of Chinese-speaking people, subscale scores range from 1-6, with a higher score indicating a higher level of positive/negative emotion

CONTACTS AND LOCATIONS:
Overall Officials: Jiayan Pan, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Jiayan Pan, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No